CLINICAL TRIAL: NCT06890780
Title: Zhujiang Hospital of Southern Medical University
Brief Title: Observation on the Correlation Between Serum/Fecal Isoflavones, Abundance of TMA-producing Bacteria and Serum TMAO in Hyperlipidemia and Healthy Subjects
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-099-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Hyperlipidemia
Keywords: hyperlipidemia; TMAO; gut microbes; Isoflavone
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperlipidemia population: Patients aged 18 to 70 years diagnosed with hyperlipidemia
- Healthy people: Between 18 and 70 years old; male weight ≥50.0kg, female weight ≥45.0kg; body mass index (BMI) within the range of 19.0-26.0 kg/m2 (including critical values); volunteers have no history of chronic diseases or serious diseases such as cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immune, mental, neuromuscular, gastrointestinal system within three years, and are in good overall health.

SUMMARY:
Previous studies have shown that trimethylamine N-oxide (TMAO), a gut microbiota-related metabolite, plays a significant role in the development and progression of cardiovascular disease (CVD). How to regulate the structure of gut microbiota to reduce circulating TMAO levels in the host is currently one of the hot topics in research. Diet is a major factor shaping the structure of gut microbiota. Through the exploration of dietary elements, we have found that multiple epidemiological studies suggest an inverse correlation between the intake of isoflavones and CVD, indicating that isoflavones are potential agents for the prevention and treatment of CVD. Interestingly, isoflavones have poor water solubility and low bioavailability. Several studies have confirmed interactions between isoflavones and gut microbiota, suggesting that the gut and gut microbiota are likely important therapeutic targets for isoflavones in preventing and treating CVD. Furthermore, a high-fat diet (HFD) is also an independent risk factor for CVD. Research literature indicates that HFD can disrupt both the gut and gut microbiota. As a biomarker for CVD risk, TMAO has been reported in some studies to increase in circulation following HFD intake, but the mechanisms behind this phenomenon require further exploration.

Based on the above literature, we propose a scientific hypothesis: Can isoflavones regulate gut microbiota and subsequently reduce serum TMAO levels in HFD-fed mice? This hypothesis can be further divided into three specific scientific questions:

Which isoflavones can reduce serum TMAO levels in HFD-fed mice?

Is gut microbiota the key factor through which isoflavones reduce serum TMAO levels in HFD-fed mice?

What mechanisms do these substances use to modulate gut microbiota?

ELIGIBILITY:
* Inclusion Criteria:
* Hyperlipidemia inclusion criteria:
* 18-70 years old；
* patients diagnosed with hyperlipidemia；
* Healthy people inclusion criteria:
* 18-70 years old；
* male weight ≥50.0kg, female weight ≥45.0kg; body mass index (BMI) within the range of 19.0-26.0 kg/m2 (including critical values);
* volunteers have no history of chronic diseases or serious diseases such as cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immune, mental, neuromuscular, gastrointestinal system within three years, and are in good overall health.
* Exclusion Criteria:
* Consuming dietary supplements (ω-3 fatty acids, probiotics, prebiotics, plant stanols/sterols) 1 month before the study;
* Using antibiotics, antidiarrheal drugs, statins, fibrates and other drugs within 2 months before the study;
* Drinking alcohol (> 2 cups per day);
* Hyperlipidemia patients with inflammatory bowel disease or irritable bowel syndrome and healthy people.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hyperlipidemia patients and healthy people
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum TMAO levels in two groups of hyperlipidemia and healthy subjects | 2023/01/01-2025/12/31
  Serum was collected from two groups of people, hyperlipidemia patients and healthy subjects, and serum TMAO levels were measured by LC-MS.
Determination of fecal TMA production capacity in two groups of hyperlipidemic subjects and healthy subjects | 2023/01/01-2025/12/31
  Serum was collected from two groups of people with hyperlipidemia and healthy subjects, and the fecal TMA production capacity of the two groups was determined by LC-MS. 16SrRNA sequencing was performed to identify strains with TMA production capacity.
The levels of fecal serum/fecal isoflavones in hyperlipidemic and healthy subjects were measured and their association with serum TMAO and TMA-producing strains was analyzed. | 2023/01/01-2025/12/31
  Simultaneously, we screened nutrients related to TMA-producing metabolic pathways in non-targeted metabolomics, such as isoflavones. Are they negatively correlated with these TMA-producing metabolic pathways? At the same time, targeted determinations were used to further screen isoflavones that have the potential to regulate TMA-producing bacterial communities. Through subsequent sample collection and metabolite analysis, we verified the regulatory ability of isoflavones on TMA-producing bacteria and clarified the biological mechanism behind them.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No